CLINICAL TRIAL: NCT00754975
Title: A Clinical Trial Comparing the Performance of the JACTAX LD DES With the TAXUS™ Libertè™ DES
Brief Title: JACTAX LD Drug Eluting Stent Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Labcoat, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBCT-H02-07
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): JACTAX LD DES
  Interventions: Device: JACTAX LD DES
- II (Active Comparator): TAXUS™ Libertè™ DES
  Interventions: Device: TAXUS™ Libertè™ DES

INTERVENTIONS:
Device: JACTAX LD DES — Drug Eluting Stent
  Arms: I
Device: TAXUS™ Libertè™ DES — Drug Eluting Stent
  Arms: II

SUMMARY:
Prospective, multi-center, randomized trial. A maximum of 130 patients will be enrolled, in a 2:1 ratio to receive either the JACTAX LD stent or the TAXUS™ Libertè™ stent to evaluate the efficacy of the product.

DETAILED DESCRIPTION:
The JACTAX Drug Eluting Stent has been designed to minimize the amount of polymer in contact with the vessel surface, thus potentially reducing the incidence of untoward side effects. The Juxtaposed Ablumenal Coating Process is capable of exclusive coating on the ablumenal side of pre-mounted bare metal stents. Juxtaposed Ablumenal Coating is a proprietary formulation containing a bioerodable polymer. The combination of the Juxtaposed Ablumenal Coating Process and Juxtaposed Ablumenal Coating create a unique microstructure surface, and reduces the amount of required polymer.

ELIGIBILITY:
General Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Patient with coronary artery disease, eligible for percutaneous coronary intervention (PCI)
3. Patient demonstrates a LVEF of ≥ 25%
4. Patient or legal guardian understands and agrees to comply with all specified study requirements and provides written informed consent to this effect.

Angiographic Inclusion Criteria

1. Target lesion is de novo native coronary artery lesion (i.e., a coronary lesion not previously treated)
2. The target lesion can be treated with a maximum of one stent, with adequate coverage onto the healthy tissue, as specified in visual estimate guidelines. Maximum lesion length is 20mm.
3. The reference vessel diameter is between 2.75mm and 3.5mm
4. Study lesion diameter stenosis is ≥70% (visual estimate) and <100% and a TIMI flow >1.
5. Study lesion has been successfully pre-dilated
6. Patients enrolled for treatment may demonstrate multiple lesions in target vessel. However lesions must be covered completely by one study stent.
7. Patient must have no more than two lesions requiring treatments. These lesions must be in different vessel distributions. For example, if the target lesion is in the LAD, then the non target lesion must be present in either the circumflex or RCA. The non-study lesion may not be in a branch vessel or distal to the target vessel location.
8. The non target lesion must be successfully treated prior to the treatment of the target lesion. The non target lesion must be treated with a TAXUS paclitaxel eluting stent or a bare metal stainless steel stent.

General Exclusion Criteria:

1. The patient has a life expectancy of less than 24 months due to another medical condition
2. Patient has a history of hypersensitivity to paclitaxel or structurally related compounds
3. Patient exhibits cardiogenic shock (systolic pressure <80mmHg and PCWP >20mmHg or cardiac index <1.8 liters/minute/m or intra-aortic balloon pump or intravenous inotropes are needed to maintain a systolic pressure >80mmHg) for any time within 24 hours prior to index procedure
4. Patient demonstrates evidence of acute or chronic renal dysfunction (serum creatinine >2.0 mg/dl or 177 umol/l)
5. Planned cardiac surgery procedure <= 9 months post index procedure
6. Patient demonstrates evidence of myocardial infarction (elevated CK, CKMB or Troponin) within 72 hours prior to the index procedure and/or CK >2X local lab's ULN, unless CK-MB is < 2X ULN
7. Patient exhibits acute ST segment elevation MI within 72 hours prior to the index procedure
8. CVA including stroke or TIA within previous 3 months
9. Patient demonstrates evidence of leukopenia
10. Patient demonstrates evidence of thrombocytopenia or thrombocytosis
11. Patient is contraindicated to ASA, clopidogrel or ticlopidine
12. Patient is currently taking warfarin or possibility of treatment with warfarin during the following 6 months post index procedure
13. Patient has been treated with paclitaxel or other chemotherapeutic agents within 12 months prior to planned index procedure
14. Anticipated treatment with paclitaxel or oral rapamycin during any period in the 9 months after the index procedure
15. Patient has received a drug eluting stent within 12 months prior to planned index procedure
16. Previous or planned treatment with intravascular brachytherapy in target vessel
17. Known allergy to stainless steel
18. Male or female with known intention to procreate within 3 months after the index procedure
19. Female of childbearing potential with a positive pregnancy test within 7 days before the index procedure or lactating or intends to become pregnant during the 9 months post index procedure

Angiographic Exclusion Criteria

1. Evidence of probable or definite thrombus of the study vessel, based on angiography or IVUS
2. Study lesion is totally occluded (TIMI flow <= 1)either at baseline or before predilatation
3. Study lesion or the study vessel proximal to the study lesion is moderately or severely calcified by visual estimate
4. Study lesion is ostial in location (within 3.0 mm of vessel origin)
5. Study lesion involving arterial segments with highly tortuous anatomy or where lesion is located within or distal to a > 60 degree bend in the vessel
6. Study lesion involves a bifurcation with a diseased (>50% stenotic) branch vessel >2.0 mm in diameter
7. Left main coronary artery disease (stenosis >50%) whether protected or unprotected
8. Target lesion length >20mm based on visual estimate by operator
9. Target vessel diameter >3.5mm based on visual estimate by operator
10. Target vessel diameter <2.75 mm based on visual estimate by operator
11. Pre-treatment of the target lesion (excluding predilation) with another interventional device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
MACE rate at 9 months | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, Principal Investigator — Elizabeth Hospital, Essen Germany
Locations (5):
- Germany (5):
  - Universitatsklinikum Bonn, Bonn
  - Cardiovascular Center Sankt Katharinen, Frankfurt
  - Hamburg University CardioVascular Center, Hamburg
  - HELIOS Klinikum, Siegburg
  - Krankenhaus der Barmherzigen Bruder, Trier

IPD SHARING:
Plan to Share IPD: No